CLINICAL TRIAL: NCT04581447
Title: Extending Time Without Diabetes After Bariatric Surgery: a Randomized Controlled Trial Comparing the Metformin Addition or Not to Standard Care
Brief Title: Extending Time Without Diabetes After Bariatric Surgery: a Trial Comparing the Metformin Addition or Not to Standard Care
Acronym: DiabOUT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P170901J; 2019-000312-28 (EudraCT Number); PHRCN-17-0337 (Other Grant/Funding Number: French ministry of Health)
Record Dates: First submitted 2020-09-28; First posted 2020-10-09 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Diabetes; Bariatric Surgery; Metformin
Keywords: Diabetes; Bariatric Surgery; Sleeve gastrectomy; Gastric bypass; Metformin
MeSH Terms: conditions — Diabetes Mellitus | interventions — Metformin; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metformin + Standard care (Experimental): The pharmacological treatment (Metformin) will start at dose of 850 mg once daily and, at one month, increased to 850 mg twice daily. The dosage will be adjusted if necessary because of gastrointestinal symptoms and information on dose change during follow-up will be collected Adherence to study medications will be assessed by pills count and plasmatic dosage (Metformin group).
  All participants will receive standardized lifestyle recommendations regularly during all the time of the study Lifestyle recommendations will be provided by a nutritionist/diabetologist every 6 months at each study visit and reinforced by dedicated consultations with a dietician and a physical activity coach as usually performed in each center. This follow-up will be standardized for each center and applied equally to patients of both groups.
  Ancillary study measuring metformin-induced enterohormones secretion will be performed on a subgroup of 30 patients randomized in this arm.
  Interventions: Drug: Metformin; Other: Standard Care; Dietary Supplement: Standardized meal
- Standard Care (Other): All participants will receive standardized lifestyle recommendations regularly during all the time of the study Lifestyle recommendations will be provided by a nutritionist/diabetologist every 6 months at each study visit and reinforced by dedicated consultations with a dietician and a physical activity coach as usually performed in each center. This follow-up will be standardized for each center and applied equally to patients of both groups.
  Ancillary study measuring metformin-induced enterohormones secretion will be performed on a subgroup of 30 patients randomized in this arm.
  Interventions: Other: Standard Care; Dietary Supplement: Standardized meal

INTERVENTIONS:
Drug: Metformin — Metformin will start at dose of 850 mg once daily and, at one month increased to 850 mg twice daily
  Arms: Metformin + Standard care
Other: Standard Care — Standard Care
Dietary Supplement: Standardized meal — Measurements of metformin-induced enterohormones secretion will be done after standardized meal test in a subgroup of patients (ancillary study)

SUMMARY:
This study is a randomized trial that evaluates the effect of metformin addition or not to standard care on the duration of diabetes remission after bariatric surgery.

DETAILED DESCRIPTION:
In addition to significant weight loss, several randomized control trials (RCTs) have demonstrated that bariatric surgery can reverse or at least improve type 2 diabetes (T2D). Despite the variability in study design and patient characteristics of these RCTs, there is a consistent favorable effect of surgery compared to medical treatment for weight loss, change in HbA1c, reduction in diabetes medications, remission of metabolic syndrome and improvement in quality of life. Diabetes remission rate is estimated from 15 to 45 % according to the 4 available RCT including the most used surgery (Roux-en-Y gastric bypass (RYGB) and sleeve gastrectomy (SG)) with at least three to five years of follow-up. These results mean that more than half of patients with type 2 diabetes are still or newly diagnosed with diabetic after surgery and that extending time of diabetes remission after bariatric surgery is of major concern.

No RCT has explored yet an intervention to extend diabetes remission. Apart from bariatric surgery, metformin is unequivocally recommended to treat both diabetes and pre-diabetes along with lifestyle interventions. Results of the Diabetes Prevention Program trial showed that metformin reduces diabetes incidence by 31% in obese patients with pre-diabetes. We hypothesized that metformin might extend the duration of diabetes remission after bariatric surgery.

The study is a randomized, controlled, open-labeled, multicenter trial.

Patients fulfilling the inclusion criteria and without any of the exclusion criteria will be randomized.

Patients will receive:

* Standardized care plus metformin treatment if randomized in the experimental group given for 3 years
* Standardized care alone if randomized in the reference group

Primary objective is to demonstrate that metformin increases the proportion of patients with T2D remission compared to standard care among ex-T2D patients operated of BS, after a 3-year period of treatment.

Secondary objectives are:

* To assess the proportion of patients with T2D partial or complete remission with metformin compared to standard care in ex-T2D patients operated of BS, after 1 and 2 years of treatment.
* To assess body weight and metabolic parameters in metformin group versus standard care.
* To assess tolerance, nutritional status and adherence to metformin in intervention group versus standard care.
* To assess micro and macroangiopathy at 3 years.
* To assess quality of life changes from baseline at 1, 2 and 3 years.
* To assess the accuracy of long term prediction score (i.e. prolonged remission assessed at the end of the study with the Ad-DiaRem score)
* To explore gut contribution to metformin metabolic effect by: (i) gut microbiota differences (diversity, composition and function) between metformin treated and non-treated individuals and (ii) measurements of metformin-induced enterohormones secretion

Patients are followed up every 6 months during 3 years in both arms. If diabetes is diagnosed during the follow-up (HbA1c > 6.5 %), the primary endpoint of the study is obtained meaning end of diabetes remission but patients will be still followed up to the end of protocol to monitor the secondary endpoints. When remission is over, the care defined by the protocol (ie metformin + standardized care or standardized care alone) should be stopped. In both groups, when remission is over, management of the disease has to be adapted according to physician's and patient's preference whatever the arm of randomization.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18-70 years old
* Having undergone gastric bypass or sleeve gastrectomy 12 to 36 +/-3 months before inclusion
* "ex-T2D" treated with at least one anti-diabetic drug before bariatric surgery or HbA1c ≥ 6.5 % before bariatric surgery
* HbA1C < 6.5 % at inclusion with no anti-hyperglycemic medications for the last three months
* Written consent

Exclusion Criteria:

* Known type 1 diabetes
* Pregnancy and breastfeeding
* Estimated glomerular filtration rate<44 ml/min (MDRD)
* Known intolerance to metformin
* Known contraindication to metformin:

  * Acute metabolic acidosis
  * Acute affection which could lead to renal deterioration (ex: dehydration, serious infection, shock, intravascular administration of iodinated contrast agent within the last 48 hours)
  * Acute or chronic disease which could lead to a tissue hypoxia (ex : severe cardiac insufficiency, severe respiratory insufficiency, myocardial infarction within the last 3 months, shock)
  * Hepatocellular insufficiency
  * Prothrombin ratio ≤ 50%
  * SGOT or SGPT levels ≥ 10 times the upper limits of the normal range
  * Alcohol use disorder
* Medications and medical conditions likely to confound the assessment of diabetes:

  * glucocorticoids treatment
  * renal graft
  * Cushing's syndrome
  * acromegaly
  * fasting plasma triglyceride > 600 mg/dl despite treatment
* Patient under legal protection

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2021-01-07 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with partial or complete T2D remission criteria | 3 years
  * Complete remission: HbA1c<5.7% and no anti-diabetic medications (except metformin in the experimental group).
  * Partial remission: defined as prediabetes level of glycaemia i.e. HbA1c<6.5% and no anti-diabetic medications (except metformin in the experimental group).

SECONDARY OUTCOMES:
Proportion of patients with partial or complete T2D remission criteria | 1 and 2 years
  * Complete remission: HbA1c<5.7% and no anti-diabetic medications (except metformin in the experimental group).
  * Partial remission: defined as prediabetes level of glycaemia i.e. HbA1c<6.5% and no anti-diabetic medications (except metformin in the experimental group).
Proportion of patients with strict complete T2D remission criteria | 3 years
Percentage of weight and BMI change | 1, 2 and 3 years
Fasting glycemia | 1, 2 and 3 years
  Assessment of the level of cardio-metabolic parameters associated to T2D. Fasting glycemia and insulinemia will be combined to report HOMA-IR (homeostatic model assessment - insulin resistance).
Fasting insulinemia | 1, 2 and 3 years
  Assessment of the level of cardio-metabolic parameters associated to T2D. Fasting glycemia and insulinemia will be combined to report HOMA-IR (homeostatic model assessment - insulin resistance).
Level of blood triglycerides | 1, 2 and 3 years
  Assessment of the level of cardio-metabolic parameters associated to T2D.
Level of blood HDL cholesterol | 1, 2 and 3 years
  Assessment of the level of cardio-metabolic parameters associated to T2D.
Blood pressure | 1, 2 and 3 years
  Systolic and diastolic blood pressure.
Level of blood albumin | 1, 2 and 3 years
  Level of nutritional parameters associated with BS
Level of blood hemoglobin | 1, 2 and 3 years
  Level of nutritional parameters associated with BS
Level of blood iron | 1, 2 and 3 years
  Level of nutritional parameters associated with BS
Level of serum ferritin | 1, 2 and 3 years
  Level of nutritional parameters associated with BS
Transferrin saturation percentage | 1, 2 and 3 years
  Level of nutritional parameters associated with BS
Level of blood calcium | 1, 2 and 3 years
  Level of nutritional parameters associated with BS
Level of blood vitamin D | 1, 2 and 3 years
  Level of nutritional parameters associated with BS
Level of blood vitamin B1 | 1, 2 and 3 years
  Level of nutritional parameters associated with BS
Level of blood vitamin B9 | 1, 2 and 3 years
  Level of nutritional parameters associated with BS
Level of blood vitamin B12 | 1, 2 and 3 years
  Level of nutritional parameters associated with BS
Proportion of adverse effects in the intervention group compared to standard care | 3 years
Number of pills taken per patient | 1, 2 and 3 years
  Adherence level assessment in the intervention group. Compliant patients are defined as taking at least 80% of assigned study pills in the intervention group.
Level of plasmatic metformin | 1, 2 and 3 years
  Adherence level assessment in the intervention group.
Proportion of retinopathy events | 3 years
Proportion of nephropathy events | 3 years
Proportion of macroangiopathy events | 3 years
Numbers and proportions of patients with quality of life changes | 1, 2 and 3 years
  assessed by EuroQol 5 Dimensions (EQ5D) auto-questionnaire
Clinical outcome at the end of the study | 3 years
  assessed by 5-year-Advanced-Diabetes Remission (5y-Ad-DiaRem) score
Changes in fecal microbiota | 1 and 3 years
Glycemia | 6 months or 12 months; under fasting condition then 30 and 90 min after a standardized meal
Insulinemia | 6 months or 12 months; under fasting condition then 30 and 90 min after a standardized meal
Level of glucagon | 6 months or 12 months; under fasting condition then 30 and 90 min after a standardized meal
Level of GLP-1 | 6 months or 12 months; under fasting condition then 30 and 90 min after a standardized meal
Level of GLP-2 | 6 months or 12 months; under fasting condition then 30 and 90 min after a standardized meal
Level of GIP | 6 months or 12 months; under fasting condition then 30 and 90 min after a standardized meal
Level of oxyntomodulin | 6 months or 12 months; under fasting condition then 30 and 90 min after a standardized meal
Level of PYY | 6 months or 12 months; under fasting condition then 30 and 90 min after a standardized meal
Level of ghrelin | 6 months or 12 months; under fasting condition then 30 and 90 min after a standardized meal
Level of glicentin | 6 months or 12 months; under fasting condition then 30 and 90 min after a standardized meal

CONTACTS AND LOCATIONS:
Overall Officials: Claire CARETTE, MD, Principal Investigator — claire.carette@aphp.fr
Locations (16):
- France (16):
  - CHU Amiens-Picardie - hôpital Nord, Amiens
  - AP-HP - hôpital Avicenne, Bobigny
  - CHU de Bordeaux - hôpital Haut-Lévêque, Bordeaux
  - AP-HP - hôpital Ambroise-Paré, Boulogne-Billancourt
  - AP-HP - hôpital Louis-Mourier, Colombes
  - Centre hospitalier intercommunal de Créteil, Créteil
  - CHU de Lille - hôpital Claude Huriez, Lille
  - AP-HM - hôpital de la Conception, Marseille
  - AP-HM - hôpital Nord, Marseille
  - AP-HP - hôpital européen Georges-Pompidou, Paris
  - AP-HP - hôpital Bichat-Claude Bernard, Paris
  - AP-HP - hôpital de la Pitié-Salpêtrière, Paris
  - Institut Mutualiste Montsouris, Paris
  - HCL - centre hospitalier Lyon-Sud, Pierre-Bénite
  - CH de Saint-Denis - hôpital Delafontaire, Saint-Denis
  - CHU de Toulouse - hôpital Larrey, Toulouse

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie results in publication could be shared. IPD detailed in the protocol could be shared for the purpose of a metaanalysis.
Supporting Information: Study Protocol, ICF
Time Frame: Two years after the last publication
Access Criteria: Data sharing must be accepted by the sponsor and the principal investigator (PI) based on a scientific project and scientific involvement of the PI team. Collaboration will be fostered.
  Teams wishing obtain IPD must meet the sponsor and PI team to present scientifics (and commercial) purpose, IPD needed, format of data transmission, and timeframe. Technical feasibility and financial support will be discussed before mandatory contractualization. Processing of shared data must comply with European General Data Protection Regulation (GDPR).